CLINICAL TRIAL: NCT00675324
Title: Bowel Preparation With Nutritional Drinks Instead of Traditional Bowel Preparation
Brief Title: Bowel Preparation Before Colonoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The bowel was not clean when the colonoscopy was performed
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Research department, Ersta Hospital (Unknown)
Responsible Party: Principal Investigator, Ulf Gustafsson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2008/104-31/3
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: Colonoscopy; Bowel preparation; Salt and electrolyte balance; Patients undergoing colonoscopy; Complication with traditional bowel preparation; Bowel purity degree without traditional bowel preparation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Traditional bowel preparation with Laxabon
  Interventions: Drug: Laxabon
- B (Active Comparator): Bowel preparation with nutritional drinks
  Interventions: Dietary Supplement: Fresubin Energy drink

INTERVENTIONS:
Drug: Laxabon — Laxabon 4 litres, starting the day (e.m.) before the colonoscopy
  Arms: A
Dietary Supplement: Fresubin Energy drink — 30 kcal/kg*day five days before colonoscopy
  Arms: B

SUMMARY:
Bowel preparation can be a troublesome procedure for patients undergoing colonoscopy. For patients with cardio-vascular and kidney disorders it may be dangerous with traditional bowel preparation with regard to salt and electrolyte balance. This study's purpose is to find out if nutritional drinks can replace traditional bowel preparation before colonoscopy in regard to Bowel purity degree, disturbances in the salt and electrolyte balance in the nutritional group versus the group that gets traditional bowel preparation. And if the patients tolerate nutritional drinks better than traditional bowel preparation.

DETAILED DESCRIPTION:
Today colonoscopy is a standard method for examination of the colon. To correctly diagnose and give adequate therapy after colonoscopy examination it is necessary with a thoroughly done bowel preparation, i.e. the intestines should preferably be empty. The ideal preparation should not only be reliable and easy to carry out but also be done without discomfort for the patient. Unfortunately we do not today have any purgative that fulfils these criteria's.

Studies have shown that Phosforal compared to Laxabon have the same or even a better effect regarding the bowel preparation and also a higher patient tolerance. The amount of side effects with Phosforal is larger and has potentially greater medical effects for the patient. Phosforal might result in serious changes in the liquid- and salt-balance and especially patients with heart diseases and kidney dysfunctions should be restricted to use this preparation.

Laxabon, on the other hand, has not showed any side effects for changes in the salt balance, but studies have shown that up to 40% of the patients are not able to drink such a large amount as four litres. Side effects as nausea, vomiting and discomfort are common.

At Ersta hospital we have for many years done research studies on the metabolic response in connection with surgery. Patients undergoing surgery for cancer in the rectum often are prepared with energy drinks in order to receive a higher energy level before the operation. As a result of this the patients often avoid nausea and have a better intestinal function after surgery. We think that this treatment has worked well on the patients but no scientific studies have been done on these patients. As a complementary result of the treatment with nutritional drinks we have found that the colon is empty already after a short time of treatment. We have also prepared some patient for colonoscopy, that due to their primary disease not are able to use traditional purgatives, with nutritional drinks for five days combined with a local purgative on the day of the examination. The colonoscopy examination on these patients were performed without any problems. We have found no studies describing this preparation before colonoscopy.

This is a study that will find out if traditional preparation before colonoscopy could be replaced by nutritional drinks combined with local purgative on the day of the examination.

ELIGIBILITY:
Inclusion Criteria:

* men
* women
* age 18-90 years

Exclusion Criteria:

* patients under 18 years
* acute colitis
* acute ileus
* seriously dementia
* patients from other counties

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Bowel purity degree | day of coclonscopy

SECONDARY OUTCOMES:
Reduction of complications for patients with cardio- vascular and kidney diseases | day of cocloscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Gustafsson, PhD, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital,, Stockholm, Stockholm County, Sweden